CLINICAL TRIAL: NCT05633758
Title: Metolazone As Early Add On Therapy For Acute Decompensated Heart Failure (MELT-HF): A Multicenter, Randomized Controlled Trial.
Brief Title: Metolazone As Early Add On Therapy For Acute Decompensated Heart Failure
Acronym: MELT-HF
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Scripps Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-14-6311
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Metolazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOC heart failure therapy and placebo pill (Arm A) (Placebo Comparator): This group will receive all standard heart failure therapy and placebo pill.
  Interventions: Drug: Placebo
- SOC heart failure therapy with addition of metolazone (Arm B) (Active Comparator): This group will receive all standard heart failure therapy with addition of metolazone.
  Interventions: Drug: Metolazone

INTERVENTIONS:
Drug: Placebo — All patients will receive standard heart failure therapy, including but not restricted to diuretics, digoxin, angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, aldosterone antagonists, hydralazine, and/or nitrates, at the discretion of the treating physician. After informed consent is obtained, patients will be randomized 1:1 to the treatment arm or placebo arm. The first placebo dose is given within six hours of administration of first dose of intravenous diuretic. The second placebo dose is given at 24-hours after the first dose.
  Other Names: NA-placebo
  Arms: SOC heart failure therapy and placebo pill (Arm A)
Drug: Metolazone — All patients will receive standard heart failure therapy, including but not restricted to diuretics, digoxin, angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta blockers, aldosterone antagonists, hydralazine, and/or nitrates, at the discretion of the treating physician. After informed consent is obtained, patients will be randomized 1:1 to the treatment arm or placebo arm. The first dose of metolazone is given within six hours of administration of first dose of intravenous diuretic The second dose of metolazone is given 24-hours after the first dose.
  Other Names: NA-Metolazone
  Arms: SOC heart failure therapy with addition of metolazone (Arm B)

SUMMARY:
The primary objective of the study is to determine efficacy of metolazone as synergistic therapy with Lasix in patients with acute decompensated heart failure. This will be a multicenter double blinded randomized placebo- controlled pilot study of the addition of 5 mg of metolazone per day for 2 days compared to placebo in patients admitted with acute decompensated heart failure.

DETAILED DESCRIPTION:
AS DESCRIBED BY THE PRINCIPAL INVESTIGATOR (DR. HEYWOOD): The primary objective of the study is to determine efficacy of metolazone as synergistic therapy with Lasix in patients with acute decompensated heart failure. This will be a multicenter double blinded randomized placebo- controlled pilot study of the addition of 5 mg of metolazone per day for 2 days compared to placebo in patients admitted with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age at time of enrollment.
* Admitted with acute decompensated heart failure based on history, physical exam, and laboratory parameters, must include both:

  1. At least 1 symptom of either dyspnea, orthopnea, or edema.
  2. At least 1 sign of rales on auscultation, peripheral edema, ascites, or pulmonary vascular congestion on chest radiography.
* Be willing to comply with protocol-specified instructions
* Able to understand and grant informed consent.

Exclusion Criteria:

* Inability to give informed consent.
* Systolic BP < 90 mmHg
* Creatinine clearance less than 20ml/min or creatinine greater than 2.5mg/dl.
* Serum Sodium less than 128meq/L, potassium levels less than 3.5meq/L
* Known adverse reaction to metolazone
* Inability to take oral medications
* Severe Aortic Stenosis (AVA < 0.8cm³)
* History of Hypertrophic Obstructive Cardiomyopathy.
* Metastatic Carcinoma
* Severe Chronic Obstructive Pulmonary Disease (COPD), FEV < 1L
* Severe dyspnea requiring prolonged CPAP or intubation
* Moderate/Severe Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Total urinary output and negative fluid balance | 48 hours
  Total urinary output and negative fluid balance in milliliters (ml) at 48 hours following administration of first dose of intravenous diuretic.

SECONDARY OUTCOMES:
Change in weight | Day 2
  Change in weight from admission to day 2
Degree of improvement in dyspnea | 6, 12, 24, 36, and 48 hours
  Dyspnea assessed at 6, 12, 24, 36, and 48 hours with Modified Borg Scale (1-10)
All cause mortality | 30 days
  All-cause mortality at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James T Heywood, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Green Torrey Pines, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No